CLINICAL TRIAL: NCT01773421
Title: An Open-label, Dose Escalation, Pharmacodynamic, Pharmacokinetic, and Effect of Food Phase 1 Study of E7820, to Determine the Maximum Tolerated Dose Following Twice Daily Oral Administration in Subjects With Unresectable Solid Tumors
Brief Title: An Open-label, Dose Escalation, Pharmacodynamic, Pharmacokinetic, and Effect of Food Phase 1 Study of E7820 to Determine the Maximum Tolerated Dose Following Twice Daily Oral Administration in Subjects With Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7820-E044-110; 2010-023655-28 (EudraCT Number)
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2018-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — N-(3-cyano-4-methyl-1H-indol-7-yl)-3-cyanobenzene-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Experimental)
  Interventions: Drug: E7820
- Part B (Experimental)
  Interventions: Drug: E7820

INTERVENTIONS:
Drug: E7820 — FOOD EFFECT STUDY:
  Each subject (a minimum of 12 subjects) will be assigned according to a randomization code to receive a single 50 mg dose of E7820 on Day 1, either after fasting for 10 hours, or immediately after consuming a high fat breakfast. Following a 7-day washout period, the subjects will crossover and a second 50 mg dose of E7820 will be administered on Day 8.
  Arms: Part A
Drug: E7820 — MTD DETERMINATION FOR BID DOSING SCHEDULE
  The initial dose of E7820 will be 50 mg BID. If allowed by the rules for dose escalation, the dose escalations will be to 60 mg BID, 80 mg BID, and 100 mg BID.
  Arms: Part B

SUMMARY:
This study consists of two Parts. Part A (Food Effect Study) and Part B (Determination of Maximum Tolerated Dose [MTD] for twice daily [BID] Dosing).Part A will be initiated first, and Part B will be initiated after the PK results of Part A have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Histological or cytological evidence of an unresectable or refractory solid tumor.
3. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
4. Subjects with known brain metastases will be eligible under the following conditions A. Have undergone complete surgical excision and are more then 1 month post surgery with no radiographic evidence of brain disease recurrence or B. Have undergone stereotactic radio surgery (gamma knife procedure) and are more then 1 month post procedure and with no radiographic evidence of brain disease progression and C. Are asymptomatic and D. Discontinued corticosteroid treatment at least 30 days prior to Cycle 1, Day 1
5. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limits of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (in the case of liver metastases less than or equal to 5 x ULN) In case alkaline phosphatase is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND subject also is known to have bone metastases, the liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
6. Adequate renal function as evidenced by serum creatinine less than or equal to 2.0 mg/dL (177 micro-mol/L) or calculated creatinine clearance greater than or equal to 40 mL/min per the Cockcroft and Gault formula
7. Provide written informed consent.
8. Are willing and able to comply with all aspects of the protocol.
9. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, hemoglobin greater than or equal to 9 g/dL (5.5 mmol/L) and platelet count greater than or equal to 100 x 109/L.
10. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [beta-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of beta-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
11. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
12. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
13. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.

Exclusion Criteria:

1. Leptomeningeal metastases or brain metastases (except as for inclusion criteria #4).
2. Active hemoptysis (at least 2.5 mL [0.5 teaspoon] bright red blood) within 3 weeks prior to the first dose of study drug.
3. Hypersensitivity to sulfonamide derivatives.
4. Subjects who have had radiation to greater than or equal to 30% of their bone marrow.
5. Subjects who require therapeutic anti-coagulant therapy with warfarin or related vitamin K antagonists. Prophylactic doses of heparin or low molecular weight heparin or thrombin inhibitors may be used in place of warfarin.
6. Left ventricular ejection fraction less than 50% on echocardiography or MUGA scanning.
7. Anticancer therapies that have not been completed at least 28 days (42 days in the case of mitomycin C or nitrosoureas) prior to treatment with E7820 (other than surgery or treatment with a protein kinase inhibitor which must have been completed no less than one week prior to treatment with E7820).
8. Incomplete recovery from previous radiotherapy, chemotherapy, or surgery other than residual cutaneous effects or stable less than Grade 2 gastrointestinal toxicity.
9. History of an ischemic cardiac event, myocardial infarction or unstable cardiac disease within 3 months before study entry.
10. A clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolongation of QTc interval greater than 480 msec.
11. Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the subject's safety or study conduct.
12. Concurrent treatment with CYP3A4 inhibitors such as verapamil, cyclosporin, quinidine, erythromycin, mibefradil, clarithramycin and azoles.
13. Concurrent treatment with drugs known to be extensively metabolized by CYP2C9 and/or CYP2C19.
14. Chronic treatment with known inducers of CYP3A4 within four weeks of receiving treatment with E7820 other than corticosteroids (Appendix 6).
15. Subjects who have a positive test result for human immunodeficiency virus (HIV), hepatitis A, hepatitis B or hepatitis C.
16. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years.
17. History of drug or alcohol dependency or abuse within approximately the last 2 years.
18. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
19. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
20. Use of illegal recreational drugs.
21. Any medical or other condition that, in the opinion of the investigator, would preclude the subject's participation in a study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2017-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Centre Utrecht, Utrecht
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the Netherlands and United Kingdom from 30 June 2011 to 12 November 2017.
Pre-assignment Details: In Part A, a total of 18 participants were enrolled, out of which 15 participants were randomized and treated. In Part B, a total of 27 participants were enrolled, out of which 26 participants were treated.
Groups:
- Treatment Phase Part A: E7820 50 mg Fed+ E7820 50 mg Fasted: Participants received E7820 50 milligram (mg), tablet, orally, under fed condition on Day 1, followed by E7820 50 mg, tablet, orally, under fasted condition on Day 8. A washout period of 7 days was maintained between the doses.
- Treatment Phase Part A: E7820 50 mg Fasted + E7820 50 mg Fed: Participants received E7820 50 mg, tablet, orally, under fasted condition on Day 1, followed by E7820 50 mg, tablet, orally, under fed condition on Day 8. A washout period of 7 days was maintained between the doses.
- Treatment Phase Part B: E7820 50 mg: Participants received E7820 50 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles or early discontinuation.
- Treatment Phase Part B: E7820 60 mg: Participants received E7820 60 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles or early discontinuation.
- Extension Phase Part A: E7820 100 mg: Participants at the end of treatment phase (who received study drug at the time of data cutoff for the primary analysis) moved on to extension phase and received E7820 100 mg, once daily, tablet, orally, under fasted condition, during 28-day cycle until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor discontinuation of E7820 development.
- Extension Phase Part B: E7820 50 mg: Participants at the end of treatment phase (who received study drug at the time of data cutoff for the primary analysis) moved on to extension phase and received E7820 50 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor discontinuation of E7820 development.
- Extension Phase Part B: E7820 60 mg: Participants at the end of treatment phase (who received study drug at the time of data cutoff for the primary analysis) moved on to extension phase and received E7820 60 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor discontinuation of E7820 development. No participants from the treatment phase Part B: E7820 60 mg entered the extension phase.
Period: Treatment Phase
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed+ E7820 50 mg Fasted | Treatment Phase Part A: E7820 50 mg Fasted + E7820 50 mg Fed | Treatment Phase Part B: E7820 50 mg | Treatment Phase Part B: E7820 60 mg | Extension Phase Part A: E7820 100 mg | Extension Phase Part B: E7820 50 mg | Extension Phase Part B: E7820 60 mg
Started | 7 | 8 | 19 | 7 | 0 | 0 | 0
Completed | 7 | 8 | 13 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 6 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed+ E7820 50 mg Fasted | Treatment Phase Part A: E7820 50 mg Fasted + E7820 50 mg Fed | Treatment Phase Part B: E7820 50 mg | Treatment Phase Part B: E7820 60 mg | Extension Phase Part A: E7820 100 mg | Extension Phase Part B: E7820 50 mg | Extension Phase Part B: E7820 60 mg
Started | 0 | 0 | 0 | 0 | 15 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 12 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Phase Part A: E7820 50 mg Fed+ E7820 50 mg Fasted: Participants received E7820 50 mg, tablet, orally, under fed condition on Day 1, followed by E7820 50 mg, tablet, orally, under fasted condition on Day 8. A washout period of 7 days was maintained between the doses.
- Total: Total of all reporting groups
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed+ E7820 50 mg Fasted | Treatment Phase Part A: E7820 50 mg Fasted + E7820 50 mg Fed | Treatment Phase Part B: E7820 50 mg | Treatment Phase Part B: E7820 60 mg | Total
Number analyzed (Participants) | 7 | 8 | 19 | 7 | 41
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 44 years | 0 | 2 | 1 | 1 | 4
  Between 45 and 64 years | 5 | 1 | 8 | 5 | 19
  Between 65 and 74 years | 1 | 3 | 9 | 1 | 14
  Greater than (>) 74 years | 1 | 2 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 2 | 15
  Male | 3 | 5 | 13 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 19 | 7 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 8 | 19 | 7 | 40
  Black or African American | 0 | 0 | 0 | 0 | 0
  Chinese | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
ECOG Score [Count of Participants; unit: Participants] — ECOG performance status was measured on 6 point scale to assess participant's performance status, where: 0 (fully active, able to carry on all pre-disease activities without restriction); 1(restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work);2(ambulatory for >50 percent of waking hours),capable of all self-care, unable to carry out any work activities);3(capable of only limited self-care, confined to bed or chair for >50 percent of waking hours); 4(completely disabled,cannot carry on any self-care,totally confined to bed or chair);5(dead).
  Participants
    0 | 1 | 4 | 7 | 1 | 13
    1 | 5 | 4 | 12 | 5 | 26
    2 | 1 | 0 | 0 | 1 | 2
    3 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase Part A: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for E7820
Time Frame: Day 1 or 8: 0.5-48 hours
Population: The pharmacokinetic (PK) analysis set included all participants who had sufficient PK data to derive at least 1 PK parameter. Participants who were evaluable at a particular time point for this endpoint were included in the assessment.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Treatment Phase Part A: E7820 50 mg Fed: Participants received E7820 50 mg, tablet, orally, under fed condition, once on Day 1 or Day 8 in treatment phase.
- Treatment Phase Part A: E7820 50 mg Fasted: Participants received E7820 50 mg, tablet, orally, under fasted condition, once on Day 1 or Day 8 in treatment phase.
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed | Treatment Phase Part A: E7820 50 mg Fasted
Number analyzed (Participants) | 12 | 14
nanogram*hour per milliliter (ng*hr/mL) | 12500 (3510) | 11500 (3490)
Statistical Analysis 1: Comparison: Treatment Phase Part A: E7820 50 mg Fed vs Treatment Phase Part A: E7820 50 mg Fasted; Test type: Equivalence — Log-transformed pharmacokinetic parameters were fit using a mixed effects model with sequence, treatment, period and sequence as fixed effects and participant as a random effect. Geometric LS means and geometric LS mean ratio were back-transformed to obtain the treatment estimates; Geometric Least Square (LS) Mean Ratio = 1.06, 90% CI 2-sided [0.97 to 1.15]

2. Primary Outcome: Treatment Phase Part A: AUC(0-t): Area Under the Plasma Concentration- Time Curve From Time 0 to t for E7820
Time Frame: Day 1 or 8: 0.5-48 hours
Population: The PK analysis set included all participants who had sufficient PK data to derive at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed | Treatment Phase Part A: E7820 50 mg Fasted
Number analyzed (Participants) | 14 | 15
ng*hr/mL | 11200 (3680) | 10500 (3460)
Statistical Analysis 1: Comparison: Treatment Phase Part A: E7820 50 mg Fed vs Treatment Phase Part A: E7820 50 mg Fasted; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 1.11, 90% CI 2-sided [1.02 to 1.2]

3. Primary Outcome: Treatment Phase Part A: Cmax: Maximum Observed Plasma Concentration for E7820
Time Frame: Day 1 or 8: 0.5-48 hours
Population: The PK analysis set included all participants who had sufficient PK data to derive at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed | Treatment Phase Part A: E7820 50 mg Fasted
Number analyzed (Participants) | 14 | 15
nanogram per milliliter (ng/mL) | 1030 (311) | 901 (242)
Statistical Analysis 1: Comparison: Treatment Phase Part A: E7820 50 mg Fed vs Treatment Phase Part A: E7820 50 mg Fasted; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Mean Ratio = 1.13, 90% CI 2-sided [1 to 1.27]

4. Primary Outcome: Treatment Phase Part B: Maximum Tolerated Dose (MTD) of E7820 BID Dosing Schedule
Description: MTD defined as the highest dose level at which no more than 1 of 6 participants experienced a dose-limiting toxicity(DLT), with the next higher dose having at least 2 of 3 or 2 of 6 participants experiencing DLTs. DLTs were defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events(CTCAE) Version 4.03 as: Neutropenia less than(<) 0.5*10^9/liter(L) for greater than(>) 5 days; neutropenia <1*10^9/L with fever; thrombocytopenia <25*10^9/L accompanied by bleeding or thrombocytopenia <10*10^9/L; any Grade 3 or 4 nonhematological toxicity for which the study drug could not be excluded as a cause (other than nausea, vomiting or diarrhea in the absence of appropriate prophylaxis) with the following clarification: Grade 3 or 4 nonhematological laboratory abnormalities for which there was no expected clinical correlation would not be considered DLTs; treatment delay of >14 days required to recover from E7820-related toxicities.
Time Frame: Up to Cycle 6 (Cycle length =28 days)
Population: MTD was assessed in safety analysis set. The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: mg
Groups:
- Treatment Phase Part B: All Participants: Participants received E7820 50 mg or 60 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles or early discontinuation.
Arm/Group | Treatment Phase Part B: All Participants
Number analyzed (Participants) | 26
mg | 50

5. Secondary Outcome: Extension Phase Part A, and Treatment and Extension Phase Part B: Number of Participants With Best Overall Response (BOR)
Description: BOR based on RECIST 1.1 for target and non-target lesions is complete response (CR) or partial response (PR) for >4 weeks or stable disease (SD) for >5 weeks from first dose. CR: disappearance of target and non-target lesions, normalization of tumor marker level, all lymph nodes must be non- pathological in size (<10 millimeter [mm] short axis). PR: at least 30% decrease in sum of diameters (SOD) of target lesions, taking as reference the baseline SOD persistence of one or more non- target lesions and/or maintenance of tumor marker level above the normal limits. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug (Baseline) up to approximately 6.6 years
Population: The efficacy evaluable analysis set: all participants with a completed tumor assessment at Baseline (Chest, Abdomen and Pelvis scans) and at least 1 complete posttreatment tumor assessment (as per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1). Overall number of participants analyzed signifies participants evaluable for this measure.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment and Extension Phase Part B: E7820 50 mg: Participants received E7820 50 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles or early discontinuation. Participants at the end of treatment phase (who received study drug at the time of data cutoff for the primary analysis) moved on to extension phase and received E7820 50 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor discontinuation of E7820 development.
- Treatment and Extension Phase Part B: E7820 60 mg: Participants received E7820 60 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles or early discontinuation. Participants at the end of treatment phase (who received study drug at the time of data cutoff for the primary analysis) moved on to extension phase and received E7820 60 mg, BID, tablet, orally, during each 28-day cycle for up to 6 cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor discontinuation of E7820 development.
Arm/Group | Extension Phase Part A: E7820 100 mg | Treatment and Extension Phase Part B: E7820 50 mg | Treatment and Extension Phase Part B: E7820 60 mg
Number analyzed (Participants) | 13 | 18 | 5
Participants
  Complete response | 0 | 0 | 0
  Partial response | 0 | 0 | 0
  Stable disease | 3 | 12 | 2

6. Secondary Outcome: Extension Phase Part A, and Treatment and Extension Phase Part B: Duration of Response
Description: Duration of response based on RECIST 1.1 for target and non-target lesions is the time from the date of first documented confirmed CR/PR until the first documentation of confirmed progressive disease (PD) or death, whichever came first. CR: disappearance of target and non-target lesions,normalization of tumor marker level,all lymph nodes must be non-pathological in size(<10 mm short axis). PR: at least 30% decrease in SOD of target lesions,taking as reference the baseline SOD persistence of one or more non- target lesions and/or maintenance of tumor marker level above the normal limits. PD:at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions,taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From date of first documented confirmed CR/PR until date of first documentation of PD or death (approximately up to 6.6 years)
Population: Duration of response was not analyzed since no participants had best overall response of CR or PR in the study.
Arm/Group | Extension Phase Part A: E7820 100 mg | Treatment and Extension Phase Part B: E7820 50 mg | Treatment and Extension Phase Part B: E7820 60 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Extension Phase Part A, and Treatment and Extension Phase Part B: Number of Participants With Death and Progressive Disease (PD)
Description: PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions. For PD: participants with best response of PD have been reported. For Death: participants with death known to have died at any point have been reported.
Time Frame: From first dose date to the date of the first documentation of confirmed PD or death (approximately up to 6.6 years)
Population: The efficacy evaluable set. Due to lack of available summarized data, data has been presented only descriptively in terms of number of participants who were known to have died and number of who had PD.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase Part A: E7820 100 mg | Treatment and Extension Phase Part B: E7820 50 mg | Treatment and Extension Phase Part B: E7820 60 mg
Number analyzed (Participants) | 13 | 18 | 7
Participants
  Death | 11 | 14 | 5
  PD | 9 | 6 | 2

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Safety assessments consisted of monitoring and recording all AEs and SAEs; regular monitoring of hematology, clinical chemistry, and urine values; physical examinations; and regular measurement of vital signs, ECG, and multiple-gated acquisition (MUGA) scans or echocardiograms.
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug (approximately up to 6.6 years)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed | Treatment Phase Part A: E7820 50 mg Fasted | Extension Phase Part A: E7820 100 mg | Treatment and Extension Phase Part B: E7820 50 mg | Treatment and Extension Phase Part B: E7820 60 mg
Number analyzed (Participants) | 15 | 15 | 15 | 19 | 7
Participants
  TEAEs | 7 | 7 | 15 | 19 | 7
  SAEs | 0 | 1 | 5 | 10 | 6

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug (approximately up to 6.6 years)
Arm/Group | Treatment Phase Part A: E7820 50 mg Fed | Treatment Phase Part A: E7820 50 mg Fasted | Extension Phase Part A: E7820 100 mg | Treatment and Extension Phase Part B: E7820 50 mg | Treatment and Extension Phase Part B: E7820 60 mg
All-Cause Mortality (participants affected / at risk) | 11/15 | 11/15 | 11/15 | 14/19 | 5/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 5/15 | 10/19 | 6/7
Other Adverse Events (participants affected / at risk) | 7/15 | 6/15 | 14/15 | 19/19 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase Part A: E7820 50 mg Fed (N=15) | Treatment Phase Part A: E7820 50 mg Fasted (N=15) | Extension Phase Part A: E7820 100 mg (N=15) | Treatment and Extension Phase Part B: E7820 50 mg (N=19) | Treatment and Extension Phase Part B: E7820 60 mg (N=7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase Part A: E7820 50 mg Fed (N=15) | Treatment Phase Part A: E7820 50 mg Fasted (N=15) | Extension Phase Part A: E7820 100 mg (N=15) | Treatment and Extension Phase Part B: E7820 50 mg (N=19) | Treatment and Extension Phase Part B: E7820 60 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 8 (19) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (7) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 7 (11) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 10 (12) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (4) | 5 (8) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (6) | 2 (7)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 5 (7) | 10 (19) | 4 (5)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (6) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (9) | 3 (3) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (7) | 2 (5) | 1 (2)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 3 (4) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 5 (7) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 | 1 (2) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (6) | 3 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 1 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 4 (5) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (4) | 7 (7) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (5) | 2 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No